CLINICAL TRIAL: NCT00754416
Title: A Prospective, Multicentre Study Evaluating the Clinical Performance of the S.E.S Shoulder Prosthesis
Brief Title: S.E.S Shoulder Arthroplasty Data Collection
Status: Terminated | Type: Observational
Why Stopped: Product no more sold
Sponsor: Zimmer Biomet (Industry)
Collaborators: Biomet France SARL (Industry)
Responsible Party: Sponsor
Other Study IDs: BMET FR 02
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Arthritis
Keywords: Shoulder Replacement
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- S.E.S prosthesis: Consecutive series of patients with a S.E.S prosthesis.

SUMMARY:
This observational study intends to collect efficacy and safety data on S.E.S shoulder system

DETAILED DESCRIPTION:
The S.E.S.® shoulder system has been developed to provide a complete solution for all the indications for Shoulder Arthroplasty, Arthritis, Rotator Cuff Arthropathy, Proximal Humeral Fracture, minimising bone resection and restoring the natural anatomy of the patient.

ELIGIBILITY:
Inclusion Criteria:

* A pre-operative level of pain and function the same as for conventional joint replacement
* A likelihood of obtaining relief of pain and improved function
* Full skeletal maturity
* Ability to follow instructions
* Good general health for age
* Willing to return for follow-up evaluations

Exclusion Criteria:

* Glenohumeral joint infection, osteomyelitis
* Neuro-muscular complications
* Inability to co-operate with and complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive series of patients received S.E.S prostheses
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2003-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Constance and oxford Scores | 6m, 1yr, 2yr, 3yr, 4yr and 5 yr

SECONDARY OUTCOMES:
Complication | Any time
Patient Satisfaction | 6m,1yr,2yr,3yr,4yr and 5yr

CONTACTS AND LOCATIONS:
Overall Officials: Laurent BEGUIN, MD, Principal Investigator — Centre hospitalier Bellevue
Locations (12):
- De Dreef Van Zonnebos 13, Schilde, Belgium
- France (11):
  - Clinique Générale, Annecy
  - Clinique St Joseph, Chambéry
  - Centre Hospitalier Général, Dax
  - Clinique Chirurgicale Orthopédique A.D.R., Maxéville
  - Clinique St Jean, Montpellier
  - IRCOS, Paris
  - Clinique St Martin, Pessac
  - Clinique Mutualiste, Saint-Etienne
  - Polyclinique de l'Atlantique, Saint-Herblain
  - Institut A. Tzanck, Saint-Laurent-du-Var
  - Institut Calot, Saint-Laurent-du-Var